CLINICAL TRIAL: NCT01512433
Title: The Clinical Efficacy of Acupuncture as an Adjunct to Methadone Treatment Services for Heroin Addicts: A Randomized Controlled Trial
Brief Title: The Clinical Efficacy of Acupuncture as an Adjunct to Methadone Treatment Services for Heroin Addicts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Yuan-Yu Chan, Principal Investigator, China Medical University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSC 100-2320-B-039-029-MY2
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Opiate Dependence
Keywords: acupuncture; methadone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- True acupuncture (Active Comparator): True acupuncture was a real acupuncture which had been used in conventional Chinese medicine practice
  Interventions: Procedure: Ture acupuncture
- Sham acupuncture (Sham Comparator): Sham acupuncture was a procedure which mimicked the real acupuncture procedure.
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Ture acupuncture — Ture acupuncture included shenmen point in the ear cartilage ridge area without electrical stimulation and Hegu (LI 4) and Zusanli (ST 36) on both hands and legs with electrical stimulation. The frequency of stimulation alternated between 20 and 100 Hz (dense and disperse, DD) at automatic 2-second intervals. The intensities of the stimulations were increased in 1 mA increments to maximal tolerable intensity.
  Arms: True acupuncture
Procedure: Sham acupuncture — The needles on the bilateral Hegu (LI 4) and Zusanli (ST 36) were then connected to the electro-acupuncture machine with zero frequencies and amplitude."DeQi"was avoided during needling.
  Arms: Sham acupuncture

SUMMARY:
The purpose of this study is to investigate the efficacy of acupuncture therapy combined with standard methadone maintenance therapy to the heroin addicts.

DETAILED DESCRIPTION:
Methadone maintenance therapy for the treatment of heroin addicts for more than 40 years , and there are many studies confirm its effectiveness, such as reduced heroin addiction, reduced high-risk needle use, reduced criminal activity. But methadone also had side effects such as drowsiness, constipation, insomnia, nausea, vomiting, sweating and respiratory depression.Then the long-term heroin addicts may irregular to take methadone, which increase the risk of reuse heroin or other drugs. Since 1996, the World Health Organization (WHO) has classified acupuncture treatment indications, including drug abuse. The purpose of this study is to investigate the efficacy of acupuncture therapy combined with standard methadone maintenance therapy to the heroin addicts.

The study will be consisted of 60 heroin addicts and the inclusion criteria were: (1) age more then 20 years; (2) fulfilled Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition criteria for opiate dependence and had been received methadone maintenance treatment for more then one month. Subjects were excluded if they: (1) concurrent treatment with antidepressant or neuroleptic medication; (2) had taking acupuncture treatment in past 30 days; (3) had severe adverse effects or events history from receiving acupuncture treatment; (4) had any serious physical illness; (5) had a significant risk of suicide; (6) ear infection; (7) were pregnant or or a woman plan to pregnant; (8) had bleeding disorders or were taking anticoagulant drugs; (9) Human Immunodeficiency Virus (HIV) positive; (10) had epilepsy, cerebral vascular disease and brain injured history.The study used a randomized, placebo-controlled study design. Patients were randomly assigned to receive methadone with verum acupuncture condition (n = 30), methadone with sham acupuncture condition (n = 30). Treatments were offered 2 times weekly for 4 weeks. Weekly measures of methadone dosage and using the visual analog scale (VAS) to assess the craving severity for 4 weeks. Using the Short Form Health Survey (SF-36) and the Pittsburgh Sleep Quality Index (PSQI) to provide an assessment of quality of life and sleep quality over the previous 4 weeks.

The study hypothesis was acupuncture had clinical efficacy upon craving severity, life quality, reduced methadone dosage and sleep quality when provided as an adjunct to a standard methadone maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

* fulfilled Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition criteria for opiate dependence and had been received methadone maintenance treatment for more then one month.

Exclusion Criteria:

* concurrent treatment with antidepressant or neuroleptic medication
* had taking acupuncture treatment in past 30 days
* had severe adverse effects or events history from receiving acupuncture treatment
* had any serious physical illness
* had a significant risk of suicide
* ear infection
* were pregnant or or a woman plan to pregnant
* had bleeding disorders or were taking anticoagulant drugs
* Human Immunodeficiency Virus (HIV) positive
* had epilepsy, cerebral vascular disease and brain injured history.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
opioid craving | four weeks
  opioid craving scores on the Visual Analog Scale

SECONDARY OUTCOMES:
sleep quality | four weeks
  sleep quality was assessed using the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI)
life quality | four weeks
  life quality was assessed using the Taiwanese version of Short Form 36 (SF-36)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of psychiatry, Armed Forces Tao-Yuan General Hospital, No.168 Zhong-Xing Road, Taoyuan, Taiwan., Longtan, Taoyuan, Taiwan